CLINICAL TRIAL: NCT01589601
Title: Palliative Care in Heart Failure (PAL-HF)
Brief Title: Palliative Care in Heart Failure
Acronym: PAL-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00032443; R01NR013428 (NIH)
Record Dates: First submitted 2012-04-24; First posted 2012-05-02 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure; Heart Diseases; Cardiovascular Diseases
Keywords: Congestive Heart Failure; Heart Failure; Palliative Care; Palliative Medicine
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual heart failure care (No Intervention): Patients will be managed by a cardiologist-directed team with expertise in the diagnosis and treatment of heart failure. Until discharge, inpatient care will focus on symptom relief and initiation of evidence-based therapies. Additional goals of care will include treatment of co-morbidities and patient education designed to assist with self-management techniques. However, after discharge, which is where the study actually takes place, patients will only receive outpatient follow-up with a heart failure cardiologist or nurse practitioner who will focus on medication titration to evidence-based dosing, titration of diuretic therapy, assessment of compliance with medical and dietary regimens, and serial monitoring of end-organ function.
- Usual care + palliative care (Active Comparator): Patients will receive an interdisciplinary, multicomponent palliative care intervention combined with state of the art heart failure management designed to assess and manage the multiple domains of quality of life at the end of life for patients with advanced heart failure, including physical symptoms, psychosocial concerns, and spiritual concerns, and to facilitate advance care planning.
  Interventions: Behavioral: Usual heart failure care; Behavioral: Interdisciplinary palliative care

INTERVENTIONS:
Behavioral: Usual heart failure care — Usual heart failure care focused on symptom relief; assessment and management of anxiety, depression, and spiritual concerns; as well as advance care planning that includes definition of care goals, resuscitation preferences, and participation in the Outlook intervention.
  Other Names: Palliative Care; Palliative Medicine; Supportive Care
  Arms: Usual care + palliative care
Behavioral: Interdisciplinary palliative care — Interdisciplinary palliative care focused on symptom relief; assessment and management of anxiety, depression, and spiritual concerns; as well as advance care planning that includes definition of care goals, resuscitation preferences, and participation in the Outlook intervention.
  Arms: Usual care + palliative care

SUMMARY:
The primary aim of the PAL-HF trial is to assess the impact of an interdisciplinary palliative care intervention combined with usual heart failure management on health-related quality of life as measured by the Kansas City Cardiomyopathy Questionnaire and the Functional Assessment of Chronic Illness Therapy with Palliative Care Subscale.

DETAILED DESCRIPTION:
Heart failure currently affects over 5 million Americans. Symptomatic patients have a median life expectancy of less than 5 years and those with late-stage disease have 1-year mortality rates approaching 90%. Despite recent therapeutic advances that reduce morbidity and mortality, heart failure continues to cause enormous suffering. Patients with advanced disease suffer not only from the physical effects of the illness, but also from psychosocial and spiritual distress. In addition, heart failure costs more than $34 billion annually to the healthcare system and a disproportionate amount is spent on patients in the last 6 months of life when some of the treatments may be either ineffective or undesired. Selected patients are candidates for aggressive treatments such as cardiac transplantation or mechanical circulatory support, but the application of these therapies to the broader heart failure population is limited by resource scarcity and their untested usefulness in older patients with significant co-morbidities.

The progressive nature of heart failure coupled with high mortality rates and poor quality of life mandates greater attention to palliative care as a routine component of heart failure management. Patients with advanced heart failure, particularly the elderly and those with significant co-morbidities, ought to be ideal candidates for palliative care that aims to relieve suffering and improve quality of life. Yet, several challenges have limited the use of palliative care approaches in heart failure:

1. Determination of Prognosis. Several validated multivariable models have been developed to predict survival, yet considerable uncertainty remains and physicians are frequently unsure whether they are caring for a patient near or far from the end of life. Patients have an even harder time and are typically overly optimistic about their survival relative to that observed or predicted by multivariable models.
2. Timing of Implementation. This prognostic uncertainty and the highly variable disease trajectories of individual patients with heart failure pose a challenge as to when palliative care interventions ought to be implemented. The most appropriate time to introduce palliative care concepts, particularly with regard to end-of-life planning, remains undefined and is linked to patient prognosis and preferences.
3. Untested Interventions. There is limited evidence from randomized controlled trials of palliative care interventions in heart failure and the majority focus on resuscitation preferences. Further, practice guidelines from major cardiovascular societies are limited on this subject.
4. Lack of Palliative Care Training of Cardiovascular Specialists . The education of cardiovascular specialists typically excludes formalized training in the principles and practice of palliative care.

Given these limitations, a properly designed and powered study is required to determine whether a multidimensional palliative care intervention in addition to usual care improves health-related outcomes relative to usual care alone in advanced heart failure patients with a highly probable short-term mortality.

PAL-HF is prospective, controlled, unblinded, 2-arm, single-center clinical trial of approximately 200 advanced heart failure patients with >50% predicted 6-month mortality randomized to usual, state of the art heart failure care or usual care combined with the PAL-HF intervention.

Patients will be randomized in a 1:1 ratio to either of 2 treatment regimens:

* Usual advanced HF care
* Usual advanced HF care + interdisciplinary palliative care focused on symptom relief; assessment and management of anxiety, depression, and spiritual concerns; as well as advance care planning that includes definition of care goals, resuscitation preferences, and participation in the Outlook intervention.

The primary endpoint will be health-related quality of life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ) and the Functional Assessment of Chronic Illness Therapy with Palliative Care Subscale (FACIT-Pal) score at 6 months

The duration of the intervention in PAL-HF is 6 months, but patients in both groups will be followed until death, or the end of the study.

The study will be completed in both arms of the trial with a post-death interview with the caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Duke University Hospital inpatient adults
* Hospitalization for acute decompensated heart failure
* Dyspnea (shortness of breath) at rest or minimal exertion plus at least 1 sign of volume overload
* Previous heart failure hospitalization within the past 1 year
* At significant risk of dying from heart failure in the next 6 months
* Anticipated discharge from hospital with anticipated ability to return to outpatient follow-up appointments

Exclusion Criteria:

* Are not an inpatient at Duke University Hospital
* Acute coronary syndrome within 30 days
* Cardiac resynchronization therapy (CRT) within the past 3 months or current plan to implant CRT device
* Active myocarditis, constrictive pericarditis
* Severe stenotic valvular disease amenable to surgical intervention
* Anticipated heart transplant or ventricular assist device within 6 months
* Renal replacement therapy
* Non-cardiac terminal illness
* Women who are pregnant or planning to become pregnant
* Inability to comply with study protocol
* Are not proficient in the English language

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Rogers, MD, Principal Investigator — Duke University Medical Center - DCRI
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Background] Hayden D, Pauler DK, Schoenfeld D. An estimator for treatment comparisons among survivors in randomized trials. Biometrics. 2005 Mar;61(1):305-10. doi: 10.1111/j.0006-341X.2005.030227.x. PMID 15737107
- [Derived] Tobin RS, Samsky MD, Kuchibhatla M, O'Connor CM, Fiuzat M, Warraich HJ, Anstrom KJ, Granger BB, Mark DB, Tulsky JA, Rogers JG, Mentz RJ, Johnson KS. Race Differences in Quality of Life following a Palliative Care Intervention in Patients with Advanced Heart Failure: Insights from the Palliative Care in Heart Failure Trial. J Palliat Med. 2022 Feb;25(2):296-300. doi: 10.1089/jpm.2021.0220. Epub 2021 Dec 1. PMID 34851740
- [Derived] Truby LK, O'Connor C, Fiuzat M, Stebbins A, Coles A, Patel CB, Granger B, Pagidipati N, Agarwal R, Rymer J, Lowenstern A, Douglas PS, Tulsky J, Rogers JG, Mentz RJ. Sex Differences in Quality of Life and Clinical Outcomes in Patients With Advanced Heart Failure: Insights From the PAL-HF Trial. Circ Heart Fail. 2020 Apr;13(4):e006134. doi: 10.1161/CIRCHEARTFAILURE.119.006134. Epub 2020 Apr 9. PMID 32268795
- [Derived] Rogers JG, Patel CB, Mentz RJ, Granger BB, Steinhauser KE, Fiuzat M, Adams PA, Speck A, Johnson KS, Krishnamoorthy A, Yang H, Anstrom KJ, Dodson GC, Taylor DH Jr, Kirchner JL, Mark DB, O'Connor CM, Tulsky JA. Palliative Care in Heart Failure: The PAL-HF Randomized, Controlled Clinical Trial. J Am Coll Cardiol. 2017 Jul 18;70(3):331-341. doi: 10.1016/j.jacc.2017.05.030. PMID 28705314
- [Derived] Mentz RJ, Tulsky JA, Granger BB, Anstrom KJ, Adams PA, Dodson GC, Fiuzat M, Johnson KS, Patel CB, Steinhauser KE, Taylor DH Jr, O'Connor CM, Rogers JG. The palliative care in heart failure trial: rationale and design. Am Heart J. 2014 Nov;168(5):645-651.e1. doi: 10.1016/j.ahj.2014.07.018. Epub 2014 Jul 30. PMID 25440791

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The duration of the intervention in PAL-HF is 6 months but patients in both groups were followed until death or until the end of the study (approximately 3.5 years). Please see the numbers "completed" in the "Overall Study" section.
Groups:
- Usual Care + Palliative Care: Patients will receive an interdisciplinary, multicomponent palliative care intervention combined with state of the art heart failure management designed to assess and manage the multiple domains of quality of life at the end of life for patients with advanced heart failure, including physical symptoms, psychosocial concerns, and spiritual concerns, and to facilitate advance care planning.
  Usual heart failure care + interdisciplinary palliative care: Usual heart failure care + interdisciplinary palliative care focused on symptom relief; assessment and management of anxiety, depression, and spiritual concerns; as well as advance care planning that includes definition of care goals, resuscitation preferences, and participation in the Outlook intervention.
Period: Overall Study
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Started | 75 | 75
Completed | 28 | 26
Not Completed | 47 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 46
  >=65 years | 54 | 50 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (12.41) | 69.8 (13.43) | 70.8 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 38 | 71
  Male | 42 | 37 | 79
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150

OUTCOME MEASURES:

1. Primary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The primary endpoint is health-related quality of life as measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ).
  The KCCQ is a 23-item, disease-specific questionnaire scored from 0-100 with high scores representing better health status.
Time Frame: Baseline, 6 months
Population: Participants that completed the baseline and 6 month KCCQ
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 73 | 74
units on a scale
  KCCQ at Baseline | 36.1 (19.80) | 31.4 (16.37)
  KCCQ at 6 Months: number analyzed (Participants) | 41 | 40
  KCCQ at 6 Months | 63.1 (20.43) | 52.1 (25.02)
Statistical Analysis 1: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority; p = 0.1641, Mixed Models Analysis; Baseline; Mean Difference (Net) = 4.8719, 95% CI 2-sided [-2.0289 to 11.7728]
Statistical Analysis 2: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — 6 Months; p = 0.0299, Mixed Models Analysis; Mean Difference (Net) = 9.4938, 95% CI 2-sided [0.9406 to 18.0470]

2. Primary Outcome: Change in Functional Assessment of Chronic Illness Therapy - Palliative Care Scale (FACIT-Pal)
Description: The primary endpoint is health-related quality of life as measured by the FACIT-Pal.
  The FACIT-Pal is a 46-item measure of self-reported quality of life (27 general quality of life; 19 palliative care) that assesses quality of life in several domains. The range of FACIT-Pal total score is 0-184, a higher score is better.
Time Frame: Baseline, 6 months
Population: Participants who completed the baseline and 6 month FACIT-Pal.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 74 | 74
units on a scale
  FACIT-Pal at Baseline | 120.6 (27.03) | 118.0 (25.12)
  FACIT-Pal at 6 months: number analyzed (Participants) | 41 | 40
  FACIT-Pal at 6 months | 136.5 (28.64) | 125.8 (30.69)
Statistical Analysis 1: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority; p = 0.5531, Mixed Models Analysis; Baseline; Mean Difference (Net) = 2.7157, 95% CI 2-sided [-6.3054 to 11.7368]
Statistical Analysis 2: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority; p = 0.0350, Mixed Models Analysis; 6 Months; Mean Difference (Net) = 11.7730, 95% CI 2-sided [0.8409 to 22.7052]

3. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) - Depression and Anxiety
Description: Depression and anxiety will be assessed in all patients using the self-administered Hospital Anxiety and Depression Scale (HADS) at 2 weeks, 3 months, and 6 months.
  Range of HADS total score is 0-42. It is divided into depression and anxiety. Each is 0-21. A score of 11 or higher indicates the possible presence of the mood disorder (clinical caseness) with a score of 8 to 10 being suggestive of the presence of the respective state. The two subscales, anxiety and depression, have been found to be independent measures. In its current form the HADS in this study is divided into 3 ranges: normal (0-7), borderline (8-10), abnormal (11-21). Movement between categories would constitute a clinically significant change in the health status.
Time Frame: Baseline (2 weeks post hospital discharge), 3 months, 6 months
Population: Participants that completed the baseline, 3 month, and 6 month HADS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 59 | 54
units on a scale
  HADS Anxiety at 2 weeks | 5.7 (4.85) | 7.2 (4.36)
  HADS Anxiety at 3 months: number analyzed (Participants) | 46 | 43
  HADS Anxiety at 3 months | 5.0 (4.7) | 6.0 (4.16)
  HADS Anxiety at 6 months: number analyzed (Participants) | 41 | 39
  HADS Anxiety at 6 months | 3.7 (3.96) | 6.2 (4.75)
  HADS Depression at 2 weeks | 6.0 (3.90) | 7.3 (4.34)
  HADS Depression at 3 months: number analyzed (Participants) | 46 | 43
  HADS Depression at 3 months | 5.6 (4.12) | 6.3 (4.23)
  HADS Depression at 6 months: number analyzed (Participants) | 41 | 39
  HADS Depression at 6 months | 4.6 (3.63) | 6.4 (4.29)
Statistical Analysis 1: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Anxiety 2 weeks; p = 0.1592, Mixed Models Analysis; Mean Difference (Net) = -1.2436, 95% CI 2-sided [-2.9817 to 0.4945]
Statistical Analysis 2: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Anxiety 3 months; p = 0.3657, Mixed Models Analysis; Mean Difference (Net) = -0.7946, 95% CI 2-sided [-2.5285 to 0.9393]
Statistical Analysis 3: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Anxiety 6 months; p = 0.0480, Mixed Models Analysis; Mean Difference (Net) = -1.8269, 95% CI 2-sided [-3.6375 to -0.0164]
Statistical Analysis 4: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Depression at 2 weeks; p = 0.2372, Mixed Models Analysis; Mean Difference (Net) = -0.9097, 95% CI 2-sided [-2.4253 to 0.6058]
Statistical Analysis 5: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Depression 3 months; p = 0.4237, Mixed Models Analysis; Mean Difference (Net) = -0.6592, 95% CI 2-sided [-2.2862 to 0.9678]
Statistical Analysis 6: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — HADS Depression at 6 months; p = 0.0202, Mixed Models Analysis; Mean Difference (Net) = -1.9379, 95% CI 2-sided [-3.5672 to -0.3085]

4. Secondary Outcome: After-Death Bereaved Family Member Interview - Hospice Version
Description: A structured interview with the caregiver of those subjects that die during the study will be conducted 6 weeks following the study subject's death using the After-Death Bereaved Family Member Interview - Hospice Version. The interview provides an assessment of patient-focused, family-centered care and assesses overall quality of care received. An overall rating is derived from the ratings questions. The scoring is calculated using a pre-formatted Microsoft Excel spreadsheet for data entry and analysis. For scoring, the 5 rating questions were summed and the final scale varied between 0 (indicating worst possible care) to 50 (best possible care).
Time Frame: 6 weeks after patient's death
Population: Overall rating scale 6 weeks after patient's death.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 21 | 26
units on a scale | 9.50 (0.548) | 8.87 (2.078)

5. Secondary Outcome: Change in FACIT-Sp
Description: Spiritual well-being will be assessed using the Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale (FACIT-Sp) at 2 weeks, 3 months, and 6 months. The FACIT-Sp is a 12 item scale which assesses the role of faith in illness and meaning, peace, and purpose in life. The range of FACIT-Sp 12 score is 0-48, with higher values representing an increased spirituality across the range of religious traditions.
Time Frame: Baseline (2 weeks post hospital discharge), 3 months, 6 months
Population: Participants that completed the baseline, 3 month, and 6 month FACIT-Sp.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 57 | 55
units on a scale
  FACIT-Sp at 2 weeks | 36.4 (9.62) | 35.3 (8.75)
  FACIT-Sp at 3 months: number analyzed (Participants) | 46 | 43
  FACIT-Sp at 3 months | 37.1 (9.98) | 35.9 (9.77)
  FACIT-Sp at 6 months: number analyzed (Participants) | 41 | 38
  FACIT-Sp at 6 months | 39.6 (8.08) | 35.5 (10.27)
Statistical Analysis 1: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — FACIT-Sp at 2 weeks; p = 0.5857, Mixed Models Analysis; Mean Difference (Net) = 0.9413, 95% CI 2-sided [-2.4666 to 4.3493]
Statistical Analysis 2: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — FACIT-Sp at 3 months; p = 0.5655, Mixed Models Analysis; Mean Difference (Net) = 1.1174, 95% CI 2-sided [-2.7246 to 4.9594]
Statistical Analysis 3: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — FACIT-Sp at 6 months; p = 0.0271, Mixed Models Analysis; Mean Difference (Net) = 3.9809, 95% CI 2-sided [0.4581 to 7.5036]

6. Secondary Outcome: Utilization and Cost Measured by the Aggregate Cost of Care
Description: The investigators will use administrative data from Duke Health System to estimate costs of care to determine the cost effectiveness of palliative care versus normal care. At all follow-up points in the study (2 weeks, 6 weeks, 3 months, 6 months, and every 6 months thereafter), patients will be asked if they received care outside of the Duke Health System and to estimate the number of physician visits and/or days in the hospital. The cost of such care will be estimated using the Medical Expenditure Panel Survey and included in the aggregate cost of care from randomization until completion of the study.
  Due to administrative delays, constraints and time to access the cost data, the study team is still working through the data aggregation for full utilization comparison as well as cost comparison.
Time Frame: time of randomization until end of follow-up, approximately 3.5 years
Population: Data not collected.
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Utilization and Cost Measured by Hospital Readmissions
Description: We evaluated the total burden of all-cause, cardiovascular and Heart Failure-specific readmissions with the palliative care intervention compared to usual care.
Time Frame: Baseline (2 weeks post hospital discharge), 6 months
Measure: Number; unit: Number of readmissions
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
Number analyzed (Participants) | 75 | 75
Number of readmissions
  All-cause readmissions | 61 | 69
  Cardiosvascular readmissions | 50 | 47
  Heart failure readmissions | 36 | 35
  Non-Cardiovascular readmissions | 11 | 22
Statistical Analysis 1: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — All-cause readmissions, Poisson regression with log link and Pearson scale; p = 0.56, Poisson regression
Statistical Analysis 2: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — Cardiovascular readmissions, Poisson regression with log link and Pearson scale; p = 0.80, Poisson regression
Statistical Analysis 3: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — Heart failure readmissions, Poisson regression with log link and Pearson scale; p = 0.92, Poisson regression
Statistical Analysis 4: Comparison: Usual Care + Palliative Care vs Usual Heart Failure Care; Test type: Superiority — Non-cardiovascular readmissions, Poisson regression with log link and Pearson scale; p = 0.12, Poisson regression

ADVERSE EVENTS:
Description: Per IRB approved protocol adverse events that required MedWatch reporting were the only adverse events collected.
Arm/Group | Usual Care + Palliative Care | Usual Heart Failure Care
All-Cause Mortality (participants affected / at risk) | 40/75 | 38/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No